CLINICAL TRIAL: NCT02388243
Title: The Computer-based Drug and Alcohol Training Assessment in Kenya
Acronym: eDATA K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Africa Institute of Mental and Brain Health (AFRIMEB) (Other)
Collaborators: Grand Challenges Canada (Other); University of British Columbia (Other); Nextgenu.org (Unknown); CliniX Healthcare Limited (Unknown); Presbyterian University of Eastern Africa (Unknown); Kenya Medical Training College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GMH 0092-04; RCT protocol (Other: AMHF)
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Alcohol-Related Disorders; Social Stigma; Substance-Related Disorders
Keywords: Brief intervention; Low and middle income countries (LMIC); eLearning; Screening; Capacity Building; Primary Health Care; Education, Medical; Education, Nursing; Education, Professional; Community Health Workers
MeSH Terms: conditions — Alcohol-Related Disorders; Social Stigma; Substance-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Brief Intervention in Public Clinic (Experimental): Written information after screening; 15 minutes or so brief intervention at recruitment with follow-up visit of about the same length after one month; in public clinic.
  Interventions: Behavioral: Brief Intervention in Public Clinic
- Screening results in Public Clinic (Active Comparator): Written information after screening; No brief intervention; in public clinic.
  Interventions: Behavioral: Screening Results in Public Clinic
- Brief Intervention in Private Clinic (Experimental): Written information after screening; 15 minutes or so brief intervention at recruitment with follow-up visit of about the same length after one month; in private clinic.
  Interventions: Behavioral: Brief Intervention in Private Clinic
- Screening results in Private Clinic (Active Comparator): Written information after screening; No brief intervention; in private clinic.
  Interventions: Behavioral: Screening Results in Private Clinic

INTERVENTIONS:
Behavioral: Brief Intervention in Public Clinic — The ASSIST-linked brief intervention includes a discussion, between the clinician and patient, of problem drinking and its associated adverse effects and how to address risky level of alcohol use, using motivational interviewing techniques, assess and manage any complication or co-morbidity uncovered, and request to the patient to follow-up in one month. Clinicians will also be asked to record their baseline and follow-up clinical assessment and management through clinical follow-up forms. The total brief intervention should be around 15 minutes, with a follow-up visit of about the same length a month later. This intervention in happening in a public clinic.
  Other Names: ASSIST-linked brief intervention in public clinic
  Arms: Brief Intervention in Public Clinic
Behavioral: Screening Results in Public Clinic — At each public clinic, a community health worker will ask patients presenting for consultation who are aged 18 years or older to be screened for healthy lifestyle and to receive feedback on their results. The screening will include self-reported weight and height, (for BMI calculation), level of physical activity, and the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). The inclusion of the BMI and level of physical activity is to mask the purpose of the intervention, by decreasing the focus on substance use. The community health worker will provide the results of the BMI, physical activity and the ASSIST and will offer a leaflet with further explanation about how to address problems with those lifestyles
  Other Names: Screening Results and Written Information in Public Clinic
  Arms: Screening results in Public Clinic
Behavioral: Brief Intervention in Private Clinic — The ASSIST-linked brief intervention includes a discussion, between the clinician and patient, of problem drinking and its associated adverse effects and how to address risky level of alcohol use, using motivational interviewing technics, assess and manage any complication or co-morbidity uncovered, and request to the patient to follow-up in one month. Clinicians will also be asked to record their baseline and follow-up clinical assessment and management through clinical follow-up forms. The total brief intervention should be around 15 minutes, with a follow-up visit of about the same length a month later. This intervention in happening in a private clinic.
  Other Names: ASSIST-linked brief intervention in Private Clinic
  Arms: Brief Intervention in Private Clinic
Behavioral: Screening Results in Private Clinic — At each private clinic, a support staff will ask patients presenting for consultation who are aged 18 years or older to be screened for healthy lifestyle and to receive feedback on their results. The screening will include self-reported weight and height, (for BMI calculation), level of physical activity, and the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). The inclusion of the BMI and level of physical activity is to mask the purpose of the intervention, by decreasing the focus on substance use. The support staff will provide the results of the BMI, physical activity and the ASSIST, and will offer a leaflet with further explanation about how to address problems with those lifestyles.
  Other Names: Screening Results and Written Information in Private Clinic
  Arms: Screening results in Private Clinic

SUMMARY:
The purpose of the two RCT registered here is to determine whether clinicians trained on the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST)-linked brief intervention (BI) through the NextGenU.org model of training are able to deliver effective brief intervention for risky level of alcohol use. It is one study part of a larger program of research.

The investigators hypothesize that the NextGenU.org model of online training with mentor and peer activities is an effective way to train clinicians to deliver the ASSIST-linked brief intervention. The investigators hypothesize that eligible participants receiving the brief intervention will decrease their alcohol consumption and experienced improved health and social outcomes more than those receiving only screening results and written information (p<0.05). The investigators hypothesize the level of decrease in alcohol consumption will be similar to that of trials conducted in high-income countries (HIC).

DETAILED DESCRIPTION:
The purpose of this project is to answer the challenge of integration of screening and core packages of Mental Health (MH) and Substance Use Disorder (SUD) services into routine primary health care (PHC) through innovative e-learning technologies. The training of health professionals in Kenya (and other LMIC) has very limited content on addressing alcohol, tobacco and other substance use disorder in PHC. The investigators aim to help address this problems by adapting NextGenU training model for capacity-building of health care providers in LMIC to provide SUD screening and core services in PHC. NextGenU.org draws on already-existing, free, expert-created competencies and computer-based learning resources from accredited sources to assemble courses certified by its network of partners. The computer-based didactic learning experience is complemented with 1) peer-to-peer interactions in a local and global community of learners simultaneously studying this topic, and 2) the use of local qualified mentors, which can supplement the training taking into account local variations in organizational structures, culture, tradition and beliefs.

The intervention evaluated through this program of research includes training lay health worker or facility support staff to screen patients presenting to the facility. Those support staff then refer those who are at moderate or high risk from tobacco, alcohol or other substance use to trained PHC clinician for brief intervention (BI) related to any of the substances they use at risky level. The training intervention includes teaching the clinicians to deliver BI, and identify and manage co-morbidities or complications. The program of research around that intervention includes (1) a developmental evaluation of the on-line training through a pilot with students and clinical faculties in educational institutions, followed by the assessment of the training of already practicing health care providers in the field; (2) pre and post training assessment of clinicians and non-clinicians knowledge, attitudes and skills (including assessing their level of stigma toward those who use psychoactive substances); (3) RCTs to assess the impact of the BI on alcohol consumption and other health and social variables of interest in public and private facilities; and (4) the assessment of the impact of quality improvement training on sustainability of the screening and BI. This trial registration is only for the RCTs.

Two independently powered RCTs, one in private facilities and one in public facilities, will be run. The rational to run two independently powered RCT is that other studies of PHC workers training for depression in LMIC have shown that the intervention implemented in public facilities was successful at improving patients' outcomes, while it was not in private facilities. However, since a large proportion of the population uses private facilities, the investigators did not want to exclude private facilities from participating.

The RCT with public institutions takes place in two rural counties, Machakos and Makueni, chosen as they are very similar in terms of geography and socio-demographic characteristics, and are pretty typical of rural counties in Kenya and other LMIC. They both have a population of over 700,000, with a moderate burden of substance abuse for Kenya.

The RCT with private health care institutions (CliniX and Shalom) will takes place in the Nairobi metropolitan area. The Shalom facility is technically in the County of Machakos, very close to Nairobi city limit and serving a very similar population to that of the CliniX facilities (urban middle class Kenyans who can afford private health care consultations out of pocket or who have insurance through their workplace). The RCTs will be complemented with qualitative methodologies to monitor other aspects besides the clinical effectiveness of the intervention. On-going results will be shared with stakeholders, and may result in adapted implementation of the training as the study progresses, as per the developmental evaluation methodology. The context and rationale of any changes will be documented as part of the research process, and are expected to inform the development of the innovation, including scalability.

The methodology for the RCTs is based on the methodology followed by Flemming et al in their studies on BI for alcohol. These highly-ranked studies have been included in the latest version of the Cochrane meta-analysis on brief alcohol intervention.

Eligible sites for the RCTs includes those which are offering PHC, are willing and able to participate in the training program (access to electricity, internet through cell phone networks, staff expressing interest in being trained), have a sufficient number of clinicians and support staff who have completed the training to screen and deliver BI, and are amenable to follow the research protocol. The investigators aim to enlist in the training at least 4 public facilities per district, and 4 private facilities, as there are uncertainties over how many clinics will have their staff complete the training.

At each clinic, a community health worker (in public facilities) or complementary staff (in the private clinics) will offer patients presenting for consultation who are aged 18 years or older to be screened for healthy lifestyle and to receive feedback on their results. The person performing the screening will obtain consent specifically to participate in the screening. To mask the topic of the trial at this early stage and avoid potential stigmatization of participants, the study will be presented as one about general lifestyles (as was done in the Flemming et al. studies). The screening will include self-reported weight and height, (for body mass index - BMI), level of physical activity, and the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). The inclusion of the BMI and level of physical activity is to mask the purpose of the intervention, by decreasing the focus on substance use. The lay health worker will provide the results of the BMI, physical activity and the ASSIST and will offer a leaflets with further explanation about those lifestyles. The screener will send all of those who screen to moderate risks or above from alcohol use to the research assistant (RA). The RA will offer patients to participate in the RCTs, assess eligibility, obtain consent, collect baseline data and demographic, and randomize patients to either BI or no further intervention (the patients will have already received their screening results). The RA will explain that it is a study about lifestyles, without disclosing that he is asking them to participate because of their level of risk due to alcohol. Those eligible will be randomized to either the BI or the control group separately for men and women in each site using a computer-generated allocation method. All practitioners will have both control and intervention subjects in their practice.

Those in the BI arm will be asked by the research staff to show and discussed with the clinicians their screening results. The clinician will deliver the BI for alcohol use reaching moderate or high risk level from the ASSIST as well as advice to stop the consumption of harmful levels of any substances reported by the patient. The BI should include discussion of risky level of alcohol consumption, associated adverse effects, and followed the adapted ASSIST BI steps for Kenya, which include asking the patient to come back for follow-up about a month after the BI. Clinicians will record their baseline and follow-up clinical assessment and management through clinical follow-up forms. The total BI should be around 15 minutes, with a follow-up visit of about the same length. Any further follow-up will be at the discretion of the clinician, as part of on-going PHC.

To blind the subject to the control or the intervention allocation, they will be told that the trial focuses on healthy lifestyles including weight, substance use, and exercise. The clinician and complementary health workers will not be told which of their patients are randomized in the control or intervention arm. This methodology ensures appropriate concealment and should prevent contamination. The participants in both the control and the intervention arms will be contacted for follow-up interviews at one, three and six months to assess outcomes. Sub-samples of both control and intervention subjects will be selected for participation in focus groups to seek input into their experience of using the new knowledge and skills in practice, and how it might be improved in the Kenyan context.

Those patients who are ineligible on the basis of increased acute risk will be asked to discuss their ASSIST results with their PHC provider.

The primary outcome variable of interest is difference in mean alcohol consumption (previous 7 and 14 day use measured in g/week) between subjects in the intervention group and the control group, and collected through a timeline follow-back assessment. A statistical test frequently used in this type of study is an independent samples t-test. We used the SPSS SamplePower calculator to estimate the sample size needed to achieve 80% power, with a two-tailed level of significance (alpha) of 0.05. We use the number of grams of alcohol consumed per week obtained from the 1997 Flemming trial: a mean (SD) of 137.7 (135.7) g/wk in the intervention group, and 185.5 (155.2) in the control group. The sample size needed is then n=146 in each arm. The average consumption in the Flemming trial was on the lower side, with a difference in mean reduction very similar to the other studies with adequate allocation concealment included in the Cochrane review.

The assumptions used to estimate the recruitment period needed to reach that sample size are as follows: Using a conservative estimate of number of visits per day from those 18 years old and over (30 visits for each public clinic and 55 visits for private clinic), with 10% a prevalence of moderately risky levels of alcohol use, based on a study conducted in similar PHC centres in Kenya using the ASSIST; subtracting returning patients (an average of 30%). An enrollment of 80% was assumed. This is a conservative estimate, since enrollment has reached about 95% in previous studies of drug and alcohol use or mental illness, conducted by AMHF. Based on these assumptions, about 570 patients in the public clinics and 520 in the private clinics should be enrolled in three months. Loss to follow-up is estimated at 10% at one month, another 10% at three months, and another 10% at six months. At six months of follow-up it is expected to have approximately 370 recruited patients in public clinics and 340 patients in private clinics. This would result in sufficient power to detect the expected decrease in consumption separately in the public and the private sector. If for any unforeseen reason, the estimated needed sample size is not reached in three months, the enrollment period will be extended, and still have the capacity to do a 6 months follow-up on all the recruited subjects.

The lower average effect size obtained by including all studies in the Cochrane review, despite a lack of adequate concealment or other methodological issues, is a reduction of about 33g/week. Using a two-tailed t-test, a consumption by the intervention group of 117g/week versus a consumption of 150 g/week by the control group, a SD of 120 for a 95% CI of (-53.66,-12.34) and an intention to treat sample at initial enrollment of 520 (260 in each arm), the study will have a power of 87.9% to yield a statistically significant result.

The effect size used is the average across men and women. The study is not powered to assess the separate effect on each gender, but sub-analyses estimating the effect of gender as a covariate can be done. Potential confounders and effect modifiers will be tested in multiple linear and logistic regression models depending on the distribution of the outcome variable. The longitudinal data across our four proposed time points will be analyzed using a general linear model, repeated measures technique, in order to understand the effect of variations due to groups (i.e., a between-groups effect) and due to follow-up time (i.e., a within-groups effect). An interaction term between groups and follow-up time will also be fitted. Missing data will be handled through multiple imputation techniques as necessary.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Have an Assist alcohol score of 11 to 26

Exclusion Criteria:

* Being pregnant
* Reaching a score of 27 or higher in one or more substances (other than tobacco or cannabis)
* Having attended an alcohol treatment program in the last year
* Reporting symptoms of suicide
* Having severe neurological or psychiatric impairment (such as overt psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1212 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mean Difference in alcohol consumption | one, three and six month post BI
  Difference in alcohol consumption between intervention and control (average grams/week in previous 7 and 14 day use collected through a timeline follow-back assessment.)

SECONDARY OUTCOMES:
Change from baseline in frequency of drinking | baseline, one, three, and six months
  mean change in number of days per week of drinking between various time frame, in controls and in intervention participants group.
Change from baseline in alcohol consumption | baseline, one, three, and six months
  mean change in grams of alcohol consumed per week between various time frame, in controls and in intervention participants group.
Change from baseline in frequency of binge drinking | baseline, and at one, three, and six months
  mean change in number of days of drinking more than 6 drinks for men and more than 4 drinks for women, between various time frame, in controls and in intervention participants group.
Change from baseline in stigma related to alcohol use | baseline, and at one, three, and six months
  change over time in control and in intervention group in stigma score
difference between group in stigma related to alcohol use, | baseline, and at one, three, and six months
  difference at each time point in control and in intervention group in stigma score
depression and suicidality | baseline, and at one, three, and six months
  change (over time) and difference (between group at any given time) of the beck depression score and beck suicidality score.
Perceived Quality of Life WHO Quality of Life-BREF (WHOQOL-BREF) | baseline, and at one, three, and six months
  Change over time (inside group) and differences over time (between groups) in the WHOQOL-BREF. The WHOQOL-BREF is a shorter version of the original instrument that is convenient for use in large research studies or clinical trials.
risky sexual behaviors | baseline, and at one, three, and six months
  using the time follow back methods, we will assess engagement in risky sexual behaviors and compare inside a group over time, and between group at different times

OTHER OUTCOMES:
treatment outcomes | baseline, one, three, and six months
  to assess changes over time in one group and between group at various time point of other potential treatment effects such as health services utilization, housing, involvement in criminal activities, aggressive behaviors (perpetration or victim of), employment, other substance use (amount per day in average in last 4 weeks), self reported health status (using analogue scale) for psychological health, physical health and overall quality of life, satisfaction with life, self reported general health status, self reported general mental health, self reported daily activity stress, sense of belonging to community, number of sexual partners (last month and lifetime), sexually transmitted disease dx in the past.

CONTACTS AND LOCATIONS:
Overall Officials: David M Ndetei, PhD, Principal Investigator — Africa Institute of Mental and Brain Health (AFRIMEB); Erica Frank, MD, MPH, Principal Investigator — University of British Columbia, NextGenU.org; Victoria N Mutiso, PhD, Principal Investigator — Africa Institute of Mental and Brain Health (AFRIMEB); Veronic Clair, MD, Principal Investigator — University of British Columbia
Locations (10):
- Kenya (10):
  - Kibwezi subCounty Hospital, Kibwezi, Makueni County
  - Kalii Dispensary, Makindu, Makueni County
  - Kaunguni Dispensary, Makindu, Makueni County
  - Kiboko Health Centre, Makindu, Makueni County
  - Makindu subCounty Hospital, Makindu, Makueni County
  - Kola Health Centre, Machakos
  - Machakos Level 5 Hospital, Machakos
  - Mutituni Health Centre, Machakos
  - Shalom Hospital Athi River, Machakos
  - CliniX Buruburu, Nairobi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization The global burden of disease: 2004 update. Geneva: WHO; 2008
- [Background] World Health Organization. Global health risks: mortality and burden of disease attributable to selected major risks. ISBN 978 92 4 156387 1. WHO. 2009.
- [Background] World Health Organization/Wonca Integrating Mental Health into Primary Care: a global perspective Geneva: World Health Organization, 2008
- [Background] Humeniuk RE H-ES, Ali RL, Poznyak V, Monteiro MG. The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST): Manual for Use in Primary Care. Geneva, Switzerland: World Health Organization; 2010.
- [Background] mhGAP Intervention Guide for Mental, Neurological and Substance Use Disorders in Non-Specialized Health Settings: Mental Health Gap Action Programme (mhGAP). Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138690/ PMID 23741783
- [Background] Kaner EF, Beyer F, Dickinson HO, Pienaar E, Campbell F, Schlesinger C, Heather N, Saunders J, Burnand B. Effectiveness of brief alcohol interventions in primary care populations. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD004148. doi: 10.1002/14651858.CD004148.pub3. PMID 17443541
- [Background] Ndetei DM, Khasakhala LI, Ongecha-Owuor FA, Kuria MW, Mutiso V, Kokonya DA. Prevalence of substance abuse among patients in general medical facilities in Kenya. Subst Abus. 2009 Apr-Jun;30(2):182-90. doi: 10.1080/08897070902802125. PMID 19347756
- [Background] Ndetei DM KL, Odinga A. Baseline Study: The Mental Health Situation in Kangemi informal settlement Nairobi-Kenya: BasicNeeds Kenya; 2007
- [Background] Ndetei DM KL, Omolo JO. Incentives for health worker retention in Kenya: An assessment of current practice Kenya: Africa Mental Health Foundation (AMHF), Institute of Policy Analysis and Research (IPAR), Kenya; 2008 May 2008.
- [Background] Ndetei DM KL, Ongecha FA, Kokonya D, Mutiso V, Kuria M, Odhiambo G, Akanga S. A Study of Drug Use in Five Urban Centres in Kenya. African Journal of Drug and Alcohol Studies 2008;7:10.
- [Background] Ndetei DM KL, Omolo JO. Incentives for health worker retention in Kenya. Health Systems Reporter 2009
- [Background] Ndetei DM KM, Khasakhala L, Maru HM, Mutiso V, Mwangi J. Substance Abuse and Psychiatric Co-morbidities: A Case Study of Patients at Mathari Psychiatric Hospital, Nairobi, Kenya. African Journal of Drug and Alcohol Studies 2008;7:6
- [Background] Ndetei DM, Mathai M, Khasakhala LI, Mutiso V, Mbwayo AW. University medical education in Kenya: The challenges. Med Teach. 2010;32(10):812-5. doi: 10.3109/0142159X.2010.496011. PMID 20854156
- [Background] Ndetei DM OF, Malow RM, Onyancha J, Mutiso V, Kokonya D, Khasakhala L, Odhiambo G, Rosenberg R. Next Priorities for International in Kenya: Results from Cohort study of Drug Use, HIV and HCV Patterns in Five Urban Areas. International Psychology Reporter 2006;10:3
- [Background] Ndetei DM OF, Mutiso V, Kuria M, Khasakhala LI, Kokonya DA. The challenges of human resources in mental health in Kenya. South African Psychiatry Review 2007;10:4
- [Background] Ndetei DM, Pizzo M, Khasakhala LI, Maru HM, Mutiso VN, Ongecha-Owuor FA, Kokonya DA. Perceived economic and behavioural effects of the mentally ill on their relatives in Kenya: a case study of the Mathari Hospital. Afr J Psychiatry (Johannesbg). 2009 Nov;12(4):293-9. doi: 10.4314/ajpsy.v12i4.49050. PMID 20033112
- [Background] Kuria, M. Factors associated with relapse and remission of alcohol dependent persons after community based treatment. Open Journal of Psychiatry, 3, 264-272. doi: 10.4236/ojpsych.2013.32025, 2013
- [Background] McKimm J, Jollie C, Cantillon P. ABC of learning and teaching: Web based learning. BMJ. 2003 Apr 19;326(7394):870-3. doi: 10.1136/bmj.326.7394.870. No abstract available. PMID 12702625
- [Background] Phipps R, Merisotis J. What's the Difference? A Review of Contemporary Research on the Effectiveness of Distance Learning in Higher Education Policy report: The Institute for Higher Education Policy; 1999.
- [Background] Harden RM, Hart IR. An international virtual medical school (IVIMEDS): the future for medical education? Med Teach. 2002 May;24(3):261-7. doi: 10.1080/01421590220141008. PMID 12098412
- [Background] 2005 Program Evaluation Findings Report: Massachusetts Institute of Technology, MIT OpenCourseWare; 2006 June 5, 2006.
- [Background] Kahn JG YJ, Kahn JS.
- [Background] Richwine MP, McGowan JJ. A rural virtual health sciences library project: research findings with implications for next generation library services. Bull Med Libr Assoc. 2001 Jan;89(1):37-44. PMID 11209799
- [Background] Browling A, Ebrahim S. Handbook of Health Research Methods: McGraw-Hill International; 2005.
- [Background] Fleming MF, Barry KL, Manwell LB, Johnson K, London R. Brief physician advice for problem alcohol drinkers. A randomized controlled trial in community-based primary care practices. JAMA. 1997 Apr 2;277(13):1039-45. PMID 9091691
- [Background] Lillie E KM, and Stuart H. Opening Minds at University: Results of a Contact--Based Anti-Stigma Intervention Mental Health Commission of Canada.
- [Background] Bokhar MU IA. Open Source Tools: Empowered the E-learning Pedagogy in Distance Education. International Journal of Computer Technology and Applications 2011;2:6.
- See also: Africa Mental Health Foundation webpage about the Project — http://www.africamentalhealthfoundation.org/edatak.html
- See also: NextGenU site which gives access to the online courses — http://www.nextgenu.org
- See also: the funding organisation — http://www.grandchallenges.ca/